CLINICAL TRIAL: NCT02252419
Title: Combined Effect of Preoperative Dexamethasone and Intraoperative Paracetamol on Postoperative Sore Throat for Patients Undergoing Urologic Surgery
Brief Title: Combined Effect of Dexamethasone and Paracetamol for Postoperative Sore Throat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SoreThroatParacetamol
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-09

CONDITIONS: Pharyngitis
Keywords: Postoperative Period; Anesthesia, General; Intubation, Intratracheal; Dexamethasone; Acetaminophen
MeSH Terms: conditions — Pharyngitis | interventions — Dexamethasone; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Active Comparator): Dexamethasone will be administered 30 minutes before the anesthetic induction.
  Interventions: Drug: Dexamethasone
- Dexamethasone+ Paracetamol (DP) (Experimental): Dexamethasone will be administered 30 minutes before the anesthetic induction. Paracetamol will be administered at the end of the surgery.
  Interventions: Drug: Dexamethasone; Drug: Paracetamol

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone will be administered.
Drug: Paracetamol — Paracetamol will be administered.
  Arms: Dexamethasone+ Paracetamol (DP)

SUMMARY:
The investigators want to evaluate the efficacy of the dexamethasone and paracetamol for the prevention of postoperative sore throat.

DETAILED DESCRIPTION:
The postoperative sore throat is a common complication after the general anesthesia which decreases the quality of life. Dexamethasone is known to effective for the prevention of postoperative sore throat. The combined effect of the dexamethasone and paracetamol for postoperative sore throat, however, is not investigated.

The investigators want to evaluate the efficacy of the dexamethasone and paracetamol for the prevention of postoperative sore throat.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for urologic surgery under general anesthesia
* ASA I-III

Exclusion Criteria:

* Patients with recent sore throat
* Patients with neck surgery
* Patients with anticipated difficult airway
* Patients with Mallampati grade 3
* Patients with severe cardiovascular or pulmonary disease
* Patients with allergic history to dexamethasone or paracetamol
* Patients with liver function disorder
* Patients with liver disease

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-02 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative sore throat | 1 hour postoperatively
  Postoperative sore throat after 1 hour postoperatively will be measured (0:none, 1:mild, 2:moderate, 3:severe)

SECONDARY OUTCOMES:
Postoperative sore throat degree | 0, 1, 6, 24 hour postoperatively
  Postoperative sore throat degree after 0, 1, 6, 24 hour postoperatively will be measured (11 points, 0:none, 10:worst imaginable).
Postoperative pain | 0, 1, 6, 24 hour postoperatively
  Postoperative pain after 0, 1, 6, 24 hour postoperatively will be measured (11 points, 0:none, 10:worst imaginable).
Nausea | 0, 1, 6, 24 hour postoperatively
  Nausea will be measured at 0, 1, 6 and 24 hour postoperatively.
Vomiting | 0, 1, 6, 24 hour postoperatively
  Vomiting will be measured at 0, 1, 6 and 24 hour postoperatively.
Somnolence | 0, 1, 6, 24 hour postoperatively
  Somnolence will be measured at 0, 1, 6 and 24 hour postoperatively.
Shivering | 0, 1, 6, 24 hour postoperatively
  Shivering will be measured at 0, 1, 6 and 24 hour postoperatively.
Headache | 0, 1, 6, 24 hour postoperatively
  Headache will be measured at 0, 1, 6 and 24 hour postoperatively.
Hoarseness | 0, 1, 6, 24 hour postoperatively
  Hoarseness will be measured at 0, 1, 6 and 24 hour postoperatively.
Dysphagia | 0, 1, 6, 24 hour postoperatively
  Dysphagia will be measured at 0, 1, 6 and 24 hour postoperatively.
Analgesics | 0, 1, 6, 24 hour postoperatively
  Analgesics usage will be measured at 0, 1, 6 and 24 hour postoperatively.
Postoperative sore throat | 0, 6, 24 hour postoperatively
  Postoperative sore throat after 0, 6, 24 hour postoperatively will be measured (0:none, 1:mild, 2:moderate, 3:severe)

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Pyoung Park, PhD, Principal Investigator — Seoul National University of Hospital
Locations (1):
- Seolu National University of Hospital, Seoul, South Korea